CLINICAL TRIAL: NCT00094250
Title: More Effective Exercise Modalities in Older Congestive Heart Failure Patients
Brief Title: HEARTS: Heart, Exercise, and Resistance Training Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was closed due to administrative reasons; study did not enroll any participants.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel
Other Study IDs: 1272; R01HL071567 (NIH)
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-02

CONDITIONS: Cardiovascular Diseases; Heart Failure, Congestive; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Heart Diseases

INTERVENTIONS:
Behavioral: Resistance and Aerobic Training

SUMMARY:
This study is enrolling patients with congestive heart failure (CHF). The goal of the study is to see if one of two carefully monitored exercise programs can improve the ability of these patients to function and get about their activities.

DETAILED DESCRIPTION:
BACKGROUND:

The amount of functional skeletal muscle that CHF patients are able to preserve is a major independent predictor of their ability to maintain physical function. Older patients with CHF (who make up the vast majority of CHF patients) are least able to do this. The disease is marked by a loss of aerobic muscle fibers, while aging is marked by a loss of glycolytic muscle fibers. Because the disease may be physiologically different in older CHF patients than in younger ones (due to loss of both muscle types in older CHF patients), they need different therapeutic approaches. Strategy tests aimed at increasing muscle mass through resistance strength training in systolic failure patients have been rare, small, and generally lacking older participants. The studies done among younger CHF patients have shown that both aerobic, and combination aerobic and strength training can increase work capacity, oxidative muscle activity, and glycolytic muscle strength. Additionally, combination training can improve cardiac measures, including LVEF.

DESIGN NARRATIVE:

An estimated 200 participants age 65 and older with Class II and III CHF and LVEF 20% to 40% will be included in this study. Their work capacity will be measured in watts on a cycle ergometer exercise stress test (Time 1). They will be randomized by gender, race, and disease severity into two exercise groups: 1) resistance and aerobic training (RA); and 2) aerobic training (A). Both groups will exercise three times a week for 4 months. At the end of the 4 months of training, the cycle ergometer stress test will be repeated (Time 2). By comparing changes in maximum watts achieved from Time 1 to Time 2 in each group, an assessment can be made of the effectiveness of each exercise program in improving work capacity. Secondarily, measures will be performed and compared of myocardial remodeling, leg strength, and leg muscle oxidative capacity at Time 1 and Time 2. The goal of the study is to determine the following:

1. If low resistance frequent repetition resistance training combined with aerobic training increases aerobic work capacity more than pure aerobic training.
2. If any improvement in aerobic work capacity is due to changes in muscle fiber composition, local blood flow, arterial endothelial function, or some combination.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Inclusion Criteria:

* Class II and III CHF that has been clinically stable for at least 6 months
* Systolic ejection fraction (LVEF) between 20% and 40%
* Under the care of a cardiologist who is willing to have the patient participate in the study and who will continue to follow the patient medically during his/her participation
* Willing and able to undergo the screening procedures and the 1 month observation period to determine eligibility
* Willing and able to come to the research center three times a week for 4 months to participate in an exercise program consisting of either aerobic exercise only, or aerobic exercise plus resistance training
* Able to speak and read English
* Willing to participate in the study after having the study explained to him/her and has signed an informed consent form

Exclusion Criteria:

* Eligible for a cardiac rehabilitation program under Medicare rules due to a recent acute event
* Any medical condition that would make either exercise unsafe or uncomfortable, such as symptomatic COPD, severe arthritis, severe peripheral vascular disease, unstable heart disease, uncontrolled blood pressure, or neurological conditions
* Other complicating diseases, such as severe anemia or other blood dyscrasia affecting function, chronic renal failure, progressive cancer, or unstable diabetes
* Does not otherwise meet the above inclusion criteria

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Improvement in work capacity at anaerobic threshold (measured at Month 4)

SECONDARY OUTCOMES:
Improvements in muscle oxidative capacity, as measured by near infrared spectroscopy (NIRS)
Improvements in local muscle blood flow by NIRS and plethysmography
Improvement in arterial endothelial function (all measured at Month 4)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Posner, MD, Principal Investigator — Chairman of Medicine, Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States